CLINICAL TRIAL: NCT04956263
Title: A Comparison of Postprandial Glucose After a Mixed Meal Tolerance Test, and the Metabolic Effects of Insulin Withdrawal in a Crossover Study of the Dual Systemic SGLT1 and SGLT2 Inhibitor YG1699, and the Selective SGLT2 Inhibitor Dapagliflozin in Subjects With Type 1 Diabetes
Brief Title: A Comparison of Postprandial Glucose After a MMTT, and the Metabolic Effects of Insulin Withdrawal in a Crossover Study in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Youngene Therapeutics Inc., Ltd. (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YG1699-201
Record Dates: First submitted 2021-06-15; First posted 2021-07-09 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Type1diabetes; Diabetes Mellitus
Keywords: Mixed Meal Tolerance Test; Insulin Withdrawal
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: During the No Treatment Period prior to the baseline MMTT performed on Day -2, subjects will be randomized 1:1:1:1:1:1 to one of six Treatment Sequences A/B/C, A/C/B, B/C/A, B/A/C, C/B/A or C/A/B:
  * Treatment A is YG1699 10 mg
  * Treatment B is YG1699 25 mg
  * Treatment C is dapagliflozin 10 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): YG1699 10 mg
  Interventions: Drug: YG1699
- Treatment B (Experimental): YG1699 25 mg
  Interventions: Drug: YG1699
- Treatment C (Active Comparator): Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: YG1699 — YG1699 is a novel investigational dual inhibitor of sodium-dependent glucose cotransporters, SGLT1 and SGLT2, indicated as an adjunct to diet and exercise to improve glycemic control and weight loss in adults with T2DM. A subsequent indication will be developed for YG1699 to improve glycemic control in adults with T1DM.
  The proposed dosage form is a yellow, film-coated tablet for oral administration. The proposed tablet strengths for the current clinical research are 5 mg and 25 mg. The tablets are packaged in high-density polyethylene (HDPE) bottles with HDPE caps and desiccant inserters. Each HDPE bottle contains 30 tablets of drug product.
  The study drug YG1699 is manufactured by Youngene Therapeutics Inc., Ltd., China.
  Arms: Treatment A; Treatment B
Drug: Dapagliflozin — Farxiga® is a sodium-glucose cotransporter 2 (SGLT2) inhibitor. Faxiga® is available as a film-coated tablet for oral administration containing the equivalent of 5 mg dapagliflozin as dapagliflozin propanediol and the following inactive ingredients: microcrystalline cellulose, anhydrous lactose, crospovidone, silicon dioxide, and magnesium stearate. In addition, the film coating contains the following inactive ingredients: polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc, and yellow iron oxide.
  Other Names: Farxiga
  Arms: Treatment C

SUMMARY:
This is an inpatient treatment, double-blind, randomized, 3-way crossover study in T1DM subjects using insulin pump therapy.

DETAILED DESCRIPTION:
Subjects will be randomized to one of 6 treatment sequences. The randomized study drug will be administered once daily for 7 days throughout each of 3 treatment periods. Each subject will attend an in-house baseline period, the NoTreatment period, and 3 in-house treatment periods, The Active Periods, where the same assessments will be performed. At each of the in-house periods, a MMTT will be carried out on the sixth day of dosing and an insulin withdrawal test will be carried out on the seventh day of dosing.

Postprandial glycemic excursion after a MMTT will be evaluated one day prior to an insulin withdrawal test. An insulin pumps with different modes (such as open loop/closed loop) the mode used at screening will be the mode used throughout the study. Unblinded continuous glucose monitoring (CGM) will be initiated at the start of the 7-day Baseline Period (Day -7) and discontinued at End of Treatment (Day 34).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 to ≤ 60 years of age at the time of signing the informed consent.
2. Subjects diagnosed with T1DM for ≥ 12 months.
3. Subjects who are currently using an approved insulin pump, with a stable basal insulin dose. Stable is defined as < 20% change of dose during the last 2 weeks prior to Screening.
4. HbA1c < 9.5%.
5. C-peptide after carbohydrate ingestion of < 0.3 nmol/L, with simultaneous plasma glucose > 90 mg/dL. (If necessary, subjects may consume carbohydrates to raise blood glucose over 90 mg/dL as measured by YSI prior to drawing blood for C-peptide. This may be repeated as needed to ensure C-peptide is assessed when plasma glucose concentration is > 90 mg/dL).
6. Fasting BOHB ≤ 0.6 mmol/L.
7. Body mass index (BMI) within the range ≥ 18.5 to ≤ 27.0 kg/m2.
8. Female subjects must be non-pregnant and non-lactating.
9. Females of childbearing potential must use highly effective contraceptive methods, stable at least 2 months prior to the screening. Male subjects must be surgically sterile, abstinent or if engaged in sexual relations of childbearing potential, the subject and his partner must be using acceptable methods of contraception.
10. Capable of giving signed informed consent and willing to follow study procedures and commitment to the study duration

Exclusion Criteria:

1. Subject has a diagnosis of type 2 diabetes (T2DM).
2. Subject who has acute proliferative retinopathy or maculopathy, requiring acute treatment within 3 months of Screening.
3. Subject who has ≥ 3 Level 2 or ≥ 1 Level 3 hypoglycemic events, or hypoglycemic unawareness, or had a severe hypoglycemic event (Level 3) within 1 month prior to Screening.
4. Subject who has had DKA or nonketotic hyperosmolar state within 1 month of Screening, OR ≥ 2 events of DKA or nonketotic hyperosmolar state within 6 months of Screening.
5. Subject with uncontrolled hypertension, defined as persistent blood pressure (BP) systolic or diastolic > 150/90 mmHg, or hypotension, defined as BP < 90/60 mmHg. (Subjects BP may be re-checked per site SOP)
6. Subject with any clinically significant active disease of the gastrointestinal system (peptic ulcers, severe GERD, gastroparesis, any malabsorption/motility disorders, or chronic constipation). severe gastroparesis, and/or severe neuropathy, especially autonomic neuropathy, as judged by the Investigator.
7. Subject with history of heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, coronary artery bypass graft surgery, or angioplasty, unstable angina requiring medication, transient ischemic attack, cerebral infarct, or cerebral hemorrhage.
8. Subject with presence of clinically significant ECG findings (eg, QTcF > 450 msec for males, QTcF > 470 msec for females, left bundle branch block [LBBB],cardiac arrythmia) at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results, or may present a safety issue to that particular subject.
9. Subject with history of renal disease or abnormal kidney function tests at Screening (eGFR < 60 mL/min/1.73m2 as estimated using the CKD-EPI Creatinine equation).
10. History of hereditary glucose-galactose malabsorption or primary renal glucosuria
11. Subjects with a thyroid disease, not adequately controlled. (Subjects with TSH outside of reference range due to incorrect treatment may be re-screened and included after successful treatment correction.)
12. Subject with a history of significant liver disease, transaminases (AST, ALT) ≥ 2 x upper limit normal (ULN), or total bilirubin >1.5x ULN. (Laboratory results may be re-checked once on a separate day per Investigator discretion)
13. Subject shows evidence of significant active neuropsychiatric disease, or chronic seizures, or major neurological disorders. Subjects that are stable and controlled by stable doses of selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), antipsychotics and lithium for ≥ 3 months prior to screening may be allowed based on the judgement of the investigator.
14. Subject with a history of neoplastic disease within the past 5 years, except for adequately treated non-melanomatous skin carcinoma or other malignancies which have been successfully treated ≥10 years prior to screening.
15. Subject with a previous surgical treatment for obesity (bariatric surgery, gastric banding, etc.) or any other gastrointestinal surgery that may induce malabsorption, history of bowel resection > 20 cm, or any GI procedure for weight loss (including LAP-BAND®).
16. Subject with history of any major surgery within 6 months.
17. Subject with current use of any prescribed or non-prescribed drugs (other than the allowed current treatment for T1DM).
18. Subject with a history of any serious adverse reaction or hypersensitivity to any of the investigational product components or medicinal products with similar chemical structure, a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
19. Subject with a history or positive test of hepatitis B surface antigen (HBsAg), or positive test for Hepatitis C, or presence of human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibodies.
20. Subject with history of any active infection, including Coronavirus disease (COVID-19), other than mild viral illness within 30 days prior to the first dosing. (Subjects will follow site specific COVID-19 protocols during the entire study)
21. Subjects with immunizations within 14 days prior to first dosing. Administration of coronavirus (Covid-19) vaccine within 5 days prior to first dosing or if scheduled during any in-house periods. Vaccination for COVID-19 is allowed during the study if a washout period of 5 days after vaccine administration is followed before any dosing.
22. Subject with history of alcohol abuse as judged by the Investigator within approximately 1 year. Average daily alcohol intake > 2 drinks of alcoholic beverages for men and > 1 drinks of alcoholic beverages for women. (One drink is defined as 12 fluid ounces of beer (5% alcohol), 5 fluid ounces of wine (12% alcohol) or 1.5 fluid ounces of distilled spirits (40% alcohol).

    Positive alcohol breath test at Screening and check-in.
23. Subjects with a history of smoking > 5 cigarettes per day or equivalent use of any tobacco product (e.g., nicotine patch) within 6 months prior to Screening. Subjects must be able to refrain from smoking during each in-house period.
24. Subject with a history of illicit drug abuse, including marijuana, within approximately 3 months or evidence of current use as judged by the Investigator. Positive drug test, including marijuana, at Screening and check-in.
25. Subject who participated in an investigational drug/device study within 30 days or 5 half-lives within the last dose of any study drug, whichever is longer.
26. Subjects unwilling to use study-supplied CGM throughout the study duration or to abstain from using > 1000 mg acetaminophen every 6 hours, per CGM safety information, or is unable to tolerate adhesive tape or has any unresolved adverse skin reaction in the area of the sensor placement.
27. Subject with donation or loss of > 500 mL of blood within 56 days.
28. Subject who is unwilling to adhere to the protocol requirements during the study or unwilling to cooperate, or comply with the requirements of this study, or is considered by the Investigator to be an unsuitable candidate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Concentration-time curve in plasma glucose (AUC(0-120min) ) | 6th day of treatment
  To demonstrate that either dose of YG1699 produces a lower area under the concentration-time curve in plasma glucose (AUC(0-120min) ) [mg/dL*ml] expressed as percent of No Treatment mean versus Dapagliflozin after a standardized Mixed Meal Tolerance Test (MMTT), performed on the 6th day of treatment.

SECONDARY OUTCOMES:
Objectives for MMTT | 6th day of treatment
  * To evaluate the change from the No Treatment Period versus the Active Treatment Periods in plasma glucose after the MMTT, performed on the 6th day of treatment, at 2-hour postprandial (120 minutes) of YG1699 doses versus Dapagliflozin (This endpoint may become primary endpoint after interim analysis)
  * To evaluate the change from the No Treatment Period versus the Active Treatment Periods in urinary glucose excretion (UGE) after the MMTT on the 6th day of treatment, (UGE 0-180 minutes) of YG1699 doses versus Dapagliflozin
  * To evaluate the change from the No Treatment Period versus the Active Treatment Periods in plasma glucose after the MMTT, performed on the 6th day of treatment, during 3-hour postprandial (180 minutes) at individual time points, and maximum plasma glucose of YG1699 doses versus Dapagliflozin
Objectives for Insulin Withdrawal | 7th day of treatment
  • To evaluate the increment and ratio of changes from the No Treatment Period versus the Active Treatment Periods during insulin withdrawal performed on the 7th day of treatment, in:
  * Treatment Ratios (95% CI) of the following: Serum beta-hydroxybutyrate (BOHB) , plasma glucagon , plasma glucose , plasma free fatty acids (FFA)
  * Duration of insulin withdrawal
Objectives for Insulin Requirements | over 3 days prior to the MMTT
  To evaluate the change from the No Treatment Period versus the Active Treatment Periods in basal, bolus and total daily insulin dose requirements

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lapuerta P, Urbina S, He J, Wittle A, Li C, Li T, Wang H, Hompesch M. A Randomized Crossover Trial of Mixed Meal Tolerance Test Response in People with Type 1 Diabetes on Insulin Pump Therapy and YG1699 or Dapagliflozin. Clin Pharmacol Ther. 2024 Jun;115(6):1383-1390. doi: 10.1002/cpt.3225. Epub 2024 Mar 8. PMID 38456487